CLINICAL TRIAL: NCT05373355
Title: Safety and Efficacy of TLL018 in Patients With Chronic Spontaneous Urticaria.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hangzhou Highlightll Pharmaceutical Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: TLL018-204
Record Dates: First submitted 2022-05-10; First posted 2022-05-13 (Actual); Last update posted 2024-03-01 (Actual); Status verified 2023-10

CONDITIONS: Chronic Spontaneous Urticaria
MeSH Terms: conditions — Chronic Urticaria

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Cohort 1 (Experimental): TLL018 tablets 1piece,BID
  Interventions: Drug: TLL018 tablets
- Cohort 2 (Experimental): TLL018 tablets 3pieces, BID
  Interventions: Drug: TLL018 tablets
- Cohort 3 (Placebo Comparator): TLL018 placeboes 3pieces, BID
  Interventions: Drug: TLL018 tablets

INTERVENTIONS:
Drug: TLL018 tablets — Oral tablets administered at different doses BID daily for 12 weeks.
  Other Names: TLL018 Placeboes

SUMMARY:
This study is a randomized, double-blind, placebo-controlled, multicenter clinical trial of about 36 subjects with moderate to severe Chronic Spontaneous Urticaria.

DETAILED DESCRIPTION:
Successfully screened subjects will be randomized in a ratio of 1：1：1. After a 4-week screening period (day -28-0), subjects will be randomly assigned to treatment for 12 weeks.

Clinical Urticaria Activity Score (UAS), dermatological Quality of Life Index (DLQI), physical exams and Laboratory tests will be performed at baseline, the end of weeks 4, 8 and 12 respectively.

ELIGIBILITY:
Inclusion Criteria:

* Have had a diagnosis of moderate to severe Chronic Spontaneous Urticaria for at least 6 months prior to Baseline;
* Subjects with moderate to severe Chronic Spontaneous Urticaria UAS7 score ≥16 at Baseline;
* Able and willing to give written informed consent.

Exclusion Criteria:

* Other types of Chronic Urticaria (such as Artificial urticaria, cold-contact urticaria, heat-contact urticaria etc);
* Other disease with symptoms of urticaria or angioedema, e.g., Urticaria vasculitis, color Vegetarian urticaria, erythema multiforme;
* History or symptoms of malignancy in any organ system regardless of treatment, and regardless of evidence of recurrence or metastasis;
* Any uncontrolled clinically significant laboratory abnormality that would affect interpretation of study data or the subject's participation in the study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2022-05-10 (Actual); Primary Completion 2023-09-07 (Actual); Study Completion 2023-09-07 (Actual)

PRIMARY OUTCOMES:
treatment-emergent adverse events (AEs), serious adverse events (SAEs) and discontinuation due to AEs/SAEs | From day 1 to Weeks 4
  Number of participants with treatment-emergent adverse events (AEs), serious adverse events (SAEs) and discontinuation due to AEs/SAEs
adverse events (AEs) according to severity | From day 1 to Weeks 4
  Number of adverse events (AEs) according to severity
blood pressure from baseline | From day 1 to Weeks 4
  Change of blood pressure from baseline
pulse rate from baseline | From day 1 to Weeks 4
  Change of pulse rate from baseline
respiratory rate from baseline | From day 1 to Weeks 4
  Change of respiratory rate from baseline
temperature from baseline | From day 1 to Weeks 4
  Change of oral temperature from baseline
clinical laboratory abnormalities compared to baseline | From day 1 to Weeks 4
  Number of participants with clinical laboratory abnormalities compared to baseline
ECG parameters from baseline | From day 1 to Weeks 4
  Change in 12-lead electrocardiogram (ECG) parameters (PR Interval, QRS Complex, QT Interval, QTC Interval) from baseline
physical examination findings from baseline | From day 1 to Weeks 4
  Number of participants with changes in physical examination findings from baseline
Cmax of TLL018 | 0 hour (pre-dose - within 30 minutes prior to dosing), and at 0.5, 1, 2, 4 and 8 hours post-dose
  Maximum observed plasma concentration (Cmax) of TLL018

SECONDARY OUTCOMES:
treatment-emergent adverse events (AEs), serious adverse events (SAEs) and discontinuation due to AEs/SAEs | From week 4 to Weeks 12
  Number of participants with treatment-emergent adverse events (AEs), serious adverse events (SAEs) and discontinuation due to AEs/SAEs
adverse events (AEs) according to severity | From week 4 to Weeks 12
  Number of adverse events (AEs) according to severity
blood pressure from baseline | From week 4 to Weeks 12
  Change of blood pressure from baseline
pulse rate from baseline | From week 4 to Weeks 12
  Change of pulse rate from baseline
respiratory rate from baseline | From week 4 to Weeks 12
  Change of respiratory rate from baseline
temperature from baseline | From week 4 to Weeks 12
  Change of oral temperature from baseline
clinical laboratory abnormalities compared to baseline | From week 4 to Weeks 12
  Number of participants with clinical laboratory abnormalities compared to baseline
ECG parameters from baseline | From week 4 to Weeks 12
  Change in 12-lead electrocardiogram (ECG) parameters (PR Interval, QRS Complex, QT Interval, QTC Interval) from baseline
physical examination findings from baseline | From week 4 to Weeks 12
  Number of participants with changes in physical examination findings from baseline
UAS7 score decreased from baseline at week 4 | Baseline to Week 4
  Change in mean value of UAS7 score from baseline at week 4 when comparing TLL-018 with placebo
UAS7 score decreased from baseline at week 8 | Time Frame: Baseline to Week 8
  Change in mean value of UAS7 score from baseline at week 8 when comparing TLL-018 with placebo
UAS7 score decreased from baseline at week 12 | Baseline to Week 12
  Change in mean value of UAS7 score from baseline at week 12 when comparing TLL-018 with placebo
DLQI score decreased from baseline at week 4 | Baseline to Weeks 4
  Change in mean value of DLQI score from baseline at week 4 when comparing TLL-018 with placebo
DLQI score decreased from baseline at week 8 | Baseline to Weeks 8
  Change in mean value of DLQI score from baseline at week 8 when comparing TLL-018 with placebo
DLQI score decreased from baseline at week 12 | Baseline to Weeks 12
  Change in mean value of DLQI score from baseline at week 12 when comparing TLL-018 with placebo

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital For Skin Diseases,Institute of Dermatology Chinese Academy of Medical Sciences, Peking Union Medical College, Nanjing, Jiangsu, China